CLINICAL TRIAL: NCT06213545
Title: Diagnostic Accuracy of Teledermatology in Patch Test Interpretation
Acronym: Tele patch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Silada Kanokrungsee, Department of Dermatology, Siriraj hospital, Mahidol University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COA 694/2023
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Teledermatology
Keywords: teledermatology; patch test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Clinic interpretation (Experimental): After doing patch test, patient come to Siriraj hospital to interpret the results at 48 hr and 72 hr.
  Interventions: Diagnostic Test: In-clinic interpretation; Diagnostic Test: Photo interpretation
- Photo interpretation (Experimental): After doing patch test, patient take a photo to Siriraj hospital by LINE application to interpret the results at 48 hr, 72 hr and 7 days
  Interventions: Diagnostic Test: In-clinic interpretation; Diagnostic Test: Photo interpretation

INTERVENTIONS:
Diagnostic Test: In-clinic interpretation — Reading patch test result at clinic
Diagnostic Test: Photo interpretation — Reading patch test result by sending photo to clinic

SUMMARY:
The goal of this clinical trial is to learn about accuracy of teledermatology in patch test interpretation in patch test's patients population. The main question[s] it aims to answer are:

* Accuracy of teledermatology in patch test interpretation by dermatologist
* Accuracy of teledermatology in patch test interpretation by Residency
* Accuracy of teledermatology in patch test interpretation by Scitentist
* The factors influencing the interpretation of remote dermatologic patch test results from photographs of patients.

Participants will

* do patch test in Siriraj hospital and come to follow up at 48 hr and 72 hr for interpretation of patch test
* take a photo at home and sent the photo to contact clinic via online application or email on the day of 48 hr, 72 hr and 7 days following the interpretation of patch test

Researchers will compare in-clinic group and telephoto group to see if the accuracy of patch test interpretation is more or less.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study must be 18 years of age or older.
* Participants in the study must have undergone patch testing for contact allergies.
* Participants in the study should be able to take photos of test results on their back and/or arms using a mobile phone or personal camera, and send them to the researcher through the Line application and/or email within 48 hours, 96 hours, and on the 7th day.
* Participants in the study should be able to read and comprehend the questionnaire in Thai and respond to the questionnaire independently.
* Participants in the study must have at least one positive result in the patch testing.
* Participants in the study must provide consent to participate in the study by signing the informed consent document.

Exclusion Criteria:

* Participants in the study who are unable to attend follow-up appointments for result assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
grading of patch test | 48 hours, 72 hours and 7 days
  sucess, intermediate and failure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Siriraj hospital, Mahidol university, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Prohibited from laws (and/or rules,regulations,contracts), Fear of inappropriate use of data